CLINICAL TRIAL: NCT00480493
Title: STEP: Social Support To Empower Parents
Acronym: STEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Susan Sullivan-Bolyai, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R15NR008391-01 (NIH)
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent mentor contact (Experimental): Parent mentor provides face-to-face social support
  Interventions: Behavioral: STEP
- Control Arm (Active Comparator): Parent is given a phone contact
  Interventions: Behavioral: STEP

INTERVENTIONS:
Behavioral: STEP — Experimental: Minutes of parent mentor-parent participant interactions Control: Minutes of parent contact-parent participant interactions
  Other Names: Experimental arm: receives parent mentor support; Control arm: receives phone number of parent contact

SUMMARY:
This RCT intervention provides parental social support (informational, affirmational, and emotional) using parent mentors (experienced in the management of the chronic illness) for mothers and fathers of young children newly diagnosed with type 1 diabetes. The parent mentors provide both home visits and phone call support over the course of the first year after diagnosis. The hypothesis is that newly diagnosed parents who receive the intervention will perceive less parental concern and worry, less negative impact on the family, more perceived confidence and social support compared to those mothers and fathers not receiving the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Mothers and fathers of children 12 years and younger with type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sullivan-Bolyai, DNSc CNS RN, Principal Investigator — University of Massachusetts, Worcester, Graduate School of Nurisng
Locations (1):
- University of Massachusetts, Worcester, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers recruited from 2 pediatric diabetes clinics in NE US,randomized 1:1 to either E or C. Of 118 mothers approached, 30 declined due to hectic schedules or had enough support; 28 (24%) passive no. 60 mothers completed the consent and baseline data, randomized to either E (32) or C (28).
Groups:
- Parent Mentor Contact: Parent mentor provides face-to-face, phone and/or e-mail social support
- Control Arm: Parent in this group receives parent contact phone number that they can call for parent support
Period: Overall Study
Arm/Group | Parent Mentor Contact | Control Arm
Started | 32 | 28
Randomized | 32 | 28
Completed | 30 | 21
Not Completed | 2 | 7
Not completed — moved | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent Mentor Contact | Control Arm | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 28 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (6.5) | 36 (6) | 36 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Maternal Confidence Scale
Description: Maternal confidence in managing child with type 1 diabetes . Higher total scores (10 questions, minimum score of 0, maximum score of 50) mean a better outcome (greater maternal confidence)
Time Frame: 12 months
Population: All participants with data were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Parent Contact Control Arm: Parent contact control arm had a phone number only to call an experienced parent raising a child with type 1 diabetes to discuss support. The experienced parent contact did not initiate the contact.
- Parent Mentor Experimental Arm: Parent mentor experimental arm had an assigned experienced parent raising a child with type 1 diabetes. The experienced parent mentor contacted the parent and negotiated the intervention dose, depending on need.
Arm/Group | Parent Contact Control Arm | Parent Mentor Experimental Arm
Number analyzed (Participants) | 28 | 32
units on a scale | 38 (7) | 37 (10)
Statistical Analysis 1: Comparison: Parent Contact Control Arm vs Parent Mentor Experimental Arm; A 2 sided t-test was used to determine if the change in Confidence score was significantly different between the groups; Test type: Superiority or Other; p = 0.468, t-test, 2 sided; Mean Difference (Final Values) = 2.46, 95% CI 2-sided [-4.32 to 9.24], Standard Error of Mean 3.36 — Confidence scores were also compared using random-effect, mixed regression models to determine whether changes over time differed significantly between groups

2. Primary Outcome: Parent Concern
Description: Parent concern in managing child with type 1 diabetes. Higher total scores (58 questions, minimum score is 58; maximum score is 255) means more worry with managing child's diabetes care.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Contact Control Arm | Parent Mentor Experimental Arm
Number analyzed (Participants) | 28 | 32
units on a scale | 149 (38) | 154 (45)
Statistical Analysis 1: Comparison: Parent Contact Control Arm vs Parent Mentor Experimental Arm; A 2 sided t-test was used to determine if there were significant differences in Concern between the two groups at 12 months; Test type: Superiority or Other; p = 0.634, t-test, 2 sided; Mean Difference (Final Values) = 4.82, 95% CI 2-sided [-15.47 to 25.11], Standard Error of Mean 10.05 — Concern scores were also compared using random-effect, mixed regression models to determine whether changes over time differed significantly between groups

3. Primary Outcome: Worry
Description: Parent worry in managing child's care. Higher total scores (11 questions, minimum score is 11, maximum score is 44) indicate more parental worry
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Contact Control Arm | Parent Mentor Experimental Arm
Number analyzed (Participants) | 28 | 32
units on a scale | 27 (7) | 27 (7.5)
Statistical Analysis 1: Comparison: Parent Contact Control Arm vs Parent Mentor Experimental Arm; The difference in the Worry score at 12 months was compared between the groups using a 2 sided t-test; Test type: Superiority or Other; p = 0.430, t-test, 2 sided; Mean Difference (Final Values) = -2.48, 95% CI 2-sided [-8.76 to 3.80], Standard Error of Mean 3.12 — We also used a random-effect, mixed regression models to look for between group changes over time

ADVERSE EVENTS:
Time Frame: Adverse event data tracked for entire study (3 years).
Arm/Group | Parent Mentor Contact | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/28
Other Adverse Events (participants affected / at risk) | 0/32 | 0/28

LIMITATIONS AND CAVEATS:
We did not have enough parents recruited to look at structural equation modeling.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No